CLINICAL TRIAL: NCT05000073
Title: Influence of Socio-aesthetic Care on the Quality of Life of Hemodialysis Patients
Acronym: SocioAesthetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PP21064
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Insufficiencies
Keywords: Quality of life; renal dialysis; socio aesthetic care
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Other: dialysis and socio-aesthetic care
- Control arm (Active Comparator)
  Interventions: Other: dialysis

INTERVENTIONS:
Other: dialysis and socio-aesthetic care — dialysis and socio-aesthetic care
  Arms: Experimental Arm
Other: dialysis — dialysis
  Arms: Control arm

SUMMARY:
The report of the Epidemiological and Information Network in Nephrology counted 44,978 hemodialysis patients in France in 2017, with more than 93% of them attending 3 sessions per week.

This multi-weekly recourse to the healthcare system in the context of substitution treatment constantly reminds patients of their disease and has a strong impact on their quality of life.

The 2011 REIN quality of life report showed that the quality of life of patients with renal failure, particularly dialysis patients, is impaired, particularly in its physical and mental components. A recent comparative study (van Sandwijk et al., 2019) comparing hemodialysis patients with hematological cancer patients under chemotherapy supports these data.

The June 2013 report of the "Etats généraux du rein", an initiative of patient associations, called for the improvement of quality of life to be made a priority and for the possibility of using supportive care and complementary non-drug techniques to be proposed.

Socio-aesthetic care, defined "as the practice of aesthetic care for people who are suffering or vulnerable", has found its place in hospitals as a complementary discipline to medical care, particularly in oncology.

We believe that in order to improve the overall quality of life of hemodialysis patients, the quality of the experience of each session must be improved. In this perspective, the repetition of socio-aesthetic care performed during dialysis sessions could contribute to the overall improvement of the quality of life.

A national survey (Saghatchian et al., 2018) on the impact of socio-aesthetic care in oncology confirms the positive perception of this care among cancer patients. Two studies carried out in hemodialysis (Bullen et al., 2018; Unal & Balci Akpinar, 2016) using complementary techniques, such as acupuncture, massage, or foot reflexology, highlight an impact on sleep, fatigue and quality of life.

The experience of implementing socio-aesthetic care in our hemodialysis unit also leads us to believe that they positively influence the perception of the session, and therefore perhaps the quality of life measured with a validated scale, the KDQOL (Kidney Disease Quality Of Life).

Our research therefore focuses on the effectiveness of social and aesthetic care during hemodialysis sessions to improve the quality of life of the hemodialysis patient.

DETAILED DESCRIPTION:
Many studies have been conducted on the overall quality of life of hemodialysis patients, but our original approach is to hypothesize that the course of each dialysis session, taken individually, can influence the overall quality of life of patients.

We hypothesize that the repetition of socio-aesthetic care as supportive care during the dialysis session would be a non-drug means to improve the quality of life of hemodialysis patients and to improve the experience of the dialysis session, the overall satisfaction of the session.

This is a randomized open clinical trial, monocentric, with two parallel arms, comparing a social and esthetic care procedure performed during a session by two certified aesthetics at the usual treatment.

The target population for this study will be individuals suffering from chronic renal failure who have been undergoing hemodialysis in the Reims University Hospital for at least one month and who will be randomly assigned to one of the two groups:

* Experimental group with socio-aesthetic care: choice of the type of care (facial modeling, hand modeling or manicure) by the patient at the rate of one session per week for 4 weeks.
* Control unit with standard support

we use several validated scales:

* Assessment of the quality of life with the KDQOL
* Assessment of anxiety and depression with the HADS anxiety and HADS depression scale
* Analogous visual evaluation of overall satisfaction with the session

ELIGIBILITY:
inclusion criteria :

* 18 years of age or older;
* Suffering from chronic kidney failure
* On hemodialysis for 1 month
* Dialysed 3 times a week
* In heavy center ;
* fluent in French;
* Benefiting from a social security system;
* Agreeing to participate in the study exclusion criteria :
* Having cognitive problems hindering the comprehension of the tool.
* Under protection of justice (guardianship or curatorship).
* Patients allergic to the care products used
* Patients with additional precautions related to a high risk of cross-transmission such as emerging highly resistant bacteria, scabies, clostridium difficile, pulmonary tuberculosis.
* Patients in withdrawal from other dialysis centers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Scale of quality of life (KDQoL) | Day 0
  Quality of life is assess by using KDQoL from 0 (worse quality of life) to 100 (better quality of life)
Scale of quality of life (KDQoL) | At Month 1
  Quality of life is assess by using KDQoL from 0 (worse quality of life) to 100 (better quality of life)

SECONDARY OUTCOMES:
Scale of anxiety and depression (HADS) | Day 0
  Anxiety and Depression are assess by using HADS scales from 0 (no anxiety or no depression) to 21 (anxiety or depression )
Scale of anxiety and depression (HADS) | At Month 1
  Anxiety and Depression are assess by using HADS scales from 0 (no anxiety or no depression) to 21 (anxiety or depression )

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France